CLINICAL TRIAL: NCT07387549
Title: A Phase III, Multicentre, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Elafibranor in Adult Participants With Primary Sclerosing Cholangitis
Brief Title: A Study to Assess How Well and Safely Elafibranor Works in Adult Participants With Primary Sclerosing Cholangitis
Acronym: ELASCOPE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-60190-475; 2026-525242-29-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elafibranor 120 mg (Experimental): Participants will take 1 tablet of elafibranor 120 mg orally once daily
  Interventions: Drug: Elafibranor
- Placebo (Placebo Comparator): Participants will take 1 placebo tablet orally once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Elafibranor — Round and orange film coated tablet of 120 mg
  Other Names: IPN60190
  Arms: Elafibranor 120 mg
Other: Placebo — Round and orange film coated tablet of placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out how well and safely elafibranor works compared to placebo in adult participants with Primary sclerosing cholangitis (PSC). PSC is a rare disease that causes inflammation and scarring of the bile ducts in the liver. Over time, this can lead to liver damage and serious health problems, including the need for a liver transplant and death.

In this study, about 350 participants with large duct PSC will take part. Participants will be randomized to receive either elafibranor 120 mg once daily or a placebo (a tablet with no active medicine). The study includes a screening period, an treatment period, and a post-treatment safety follow-up.

During the study, participants will undergo routine clinical assessments, laboratory testing, imaging evaluations, and complete patient-reassessments to evaluate liver disease progression, symptoms, quality of life and safety.

Following the end of treatment, participants will complete a safety follow-up period at approximately four weeks. Participants may withdraw from the study at any time. Each participant may be in the study for several years, as the treatment period will continue until the study reaches enough health events among participants, which is expected to take about 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults participants aged 18 years or older
* Confirmed diagnosis of primary sclerosing cholangitis based on standard clinical, biochemical, and imaging criteria
* Compensated liver disease at screening
* Stable background therapy, where applicable prior to study entry
* Women of childbearing potential have to apply during the entire duration of the study a highly effective method of birth control
* Ability to provide written informed consent and comply with study procedures.

Exclusion Criteria:

- History or presence of other concomitant chronic liver disease

- History of hepatic decompensation, including: i) History of liver transplantation, current MELD 3.0 score ≥12 due to hepatic impairment.

ii) Evidence of complications of cirrhosis

* Participants with cirrhosis who are also classified as Child-Pugh B or C based on the Child Pugh score.
* History of biliary intervention within 60 days prior to the screening period, and/or presence of percutaneous drain or bile duct stent at SV.
* History of bacterial cholangitis, and/or participant on antibiotics for prophylaxis of recurrent cholangitis within 60 days prior to the SV.
* History or any current suspicion of cholangiocarcinoma or hepatocellular carcinoma
* Known malignancy or history of malignancy within the last 5 years, with the exception of local, successfully treated basal cell carcinoma or in-situ carcinoma of the uterine cervix.
* Medical conditions that may cause non-hepatic increases in ALP (e.g. Paget's disease).
* Administration of the following medications are prohibited as specified below:

  i) 3 months prior to baseline: norucholic acid, fibrates, seladelpar and glitazones.

ii) 3 months prior to baseline: cyclosporine, mycophenolate, pentoxifylline, and chronic systemic corticosteroids (except as part of management of IBD at an ongoing stable dose); potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazid, or nitrofurantoin).

* Participants who are currently participating in, plan to participate in, or have participated in an investigational drug or medical device study containing active substance within 30 days or five half-lives, whichever is longer, prior to the SV. - Participants with previous exposure to elafibranor.
* Electrocardiogram (ECG) with QT interval corrected by Fridericia's formula (QTcF) >450 msec in males or QTcF >470 msec in females for participants without bundle branch block.
* Significant renal disease,
* For female participants: known pregnancy, or has a positive serum pregnancy test, or lactating.
* Regular alcohol intake in excess of the recommended limit of 2 standard drinks per day for men or 1 standard drink per day for women
* History of alcohol abuse, or other substance abuse within 1 year prior to SV.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that contraindicates participation in the study.
* Mental instability or incompetence
* Participant has or is known to have tested positive for human immunodeficiency virus (HIV) type 1 or 2 at SV.
* Medical conditions that may diminish life expectancy to <2 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-04-14 (Estimated); Primary Completion 2031-04-30 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival | From baseline until the end of treatment (estimated up to 5 years)
  Event-free survival is defined as the time from randomisation to either adjudicated disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Percentage of participants with ALP level within the pre-defined level | From baseline to Week 48
  Difference between elafibranor and placebo in the percentage of participants with alkaline phosphatase (ALP) within the pre-defined level at Week 48.
Change from baseline in severity of a patient-reported cholestatic symptom: Pruritus | From baseline to Week 24
  Symptom will be assessed using a patient-reported outcome scale
Change from baseline in severity of a patient-reported cholestatic symptom: Fatigue | From baseline to Week 48
  Symptom will be assessed using a patient-reported outcome scale
Percentage of participants experiencing treatment-emergent adverse events (TEAEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interests (AESIs) | From baseline until the end of treatment (estimated up to 5 years)
  An Adverse event (AE) is any untoward medical occurrence, temporally associated with the use of study intervention, whether or not related to the study intervention. AESIs are AEs that may not be serious but are of special importance to a particular drug or class of drugs
Percentage of participants developing clinically significant changes in physical examination findings | From baseline until the end of treatment (estimated up to 5 years)
  The clinical significance will be graded by the investigator
Percentage of participants developing clinically significant changes in vital signs | From baseline until the end of treatment (estimated up to 5 years)
  The clinical significance will be graded by the investigator
Percentage of participants developing clinically significant changes in Electrocardiogram (ECG) readings. | From baseline until the end of treatment (estimated up to 5 years)
  The clinical significance will be graded by the investigator
Percentage of participants with clinically significant changes in laboratory parameters (blood chemistry, hematology, coagulation and urinalysis) | From baseline until the end of treatment (estimated up to 5 years)
  The clinical significance will be graded by the investigator
Percentage of participants developing cholangiocarcinoma (CCA), hepatocellular carcinoma (HCC), or colorectal cancer (CRC) | From baseline until the end of treatment (estimated up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/